CLINICAL TRIAL: NCT01669590
Title: Nutrient Regulation of Amino Acid Transporters in Aging Human Skeletal Muscle
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Micah Drummond, Ph.D., University of Utah
Other Study IDs: IRB_00050933
Record Dates: First submitted 2012-08-10; First posted 2012-08-21 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- old (60-75yr)
- young (18-35y)

SUMMARY:
The goal of the research project is to determine how aging and inactivity reduce the muscle anabolic effect of nutrients and lead to muscle and functional loss. The central hypothesis is that aging reduces mTORC1 signaling and the expression of skeletal muscle amino acid transporters in response to anabolic stimulation leading to reduced muscle adaptation to increased intracellular amino acid requirements. The investigators further hypothesize that inactivity exacerbates this effect with significant muscle and functional loss, and rehabilitation restores muscle signaling, metabolism and function to baseline values.

ELIGIBILITY:
Inclusion Criteria:

1 . Age between 18-35 and 60-75 yrs 2. Ability to sign informed consent 3. Mini-mental state exam score >26 4. Free-living, prior to admission

Exclusion Criteria:

1. Cardiac abnormalities considered exclusionary by the study physician (e.g., CHF, CAD, right-to-left shunt)
2. Uncontrolled endocrine or metabolic disease (e.g., hypo/hyperthyroidism, diabetes)
3. GFR <65 mL/min/1.73m2 or evidence of kidney disease or failure
4. Vascular disease or risk factors of peripheral atherosclerosis. (e.g., uncontrolled hypertension, obesity, diabetes, hypercholesterolemia > 250 mg/dl, claudication or evidence of venous or arterial insufficiency upon palpitation of femoral, popliteal and pedal arteries)
5. Risk of DVT including family history of thrombophilia, DVT, pulmonary emboli, myeloproliferative diseases including polycythemia (Hb>18 g/dL) or thrombocytosis (platelets>400x103/mL), and connective tissue diseases (positive lupus anticoagulant), hyperhomocysteinemia, deficiencies of factor V Leiden, proteins S and C, and antithrombin III
6. Use of anticoagulant therapy. (e.g., Coumadin, heparin)
7. Prior history of Heparin-Induced Thrombocytopenia (HIT)
8. Elevated systolic pressure >150 or a diastolic blood pressure > 100
9. Implanted electronic devices (e.g., pacemakers, electronic infusion pumps, stimulators)
10. Cancer or history of successfully treated cancer (less than 1 year) other than basal cell carcinoma
11. Currently on a weight-loss diet or body mass index > 30 kg/m2
12. Inability to abstain from smoking for duration of study
13. A history of > 20 pack per year smoking
14. HIV or hepatitis B or C*
15. Recent anabolic or corticosteroids use (within 3 months)
16. Subjects with hemoglobin or hematocrit lower than accepted lab values
17. Agitation/aggression disorder (by psychiatric history and exam)
18. History of stroke with motor disability
19. A recent history (<12 months) of GI bleed
20. Pregnancy as determined by a pregnancy test
21. Depression [>5 on the 15 items Geriatric Depression Scale (GDS)]
22. Alcohol or drug abuse
23. Exercise training (>1 session of moderate to high intensity aerobic or resistance exercise/week)
24. Liver disease (AST/ALT 2 times above the normal limit, hyperbilirubinemia)
25. Respiratory disease (acute upper respiratory infection, history of chronic lung disease with resting oxygen saturation <97% on room air)
26. Any other condition or event considered exclusionary by the PI and faculty physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: young and older healthy humans
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
amino acid transporter | before and after (1 and 3h) amino acid ingestion. These samples will be taken before bed rest and 7 days after bed rest.
  Muscle biopsies will be sampled from the vastus laterals before amino acid ingestion and then 1 and 3h after amino acid ingestion. Muscle biopsies will be processed using western blotting and gene expression to assess the expression of specific amino acid transporters. The investigators are interested in the change in expression of amino acid transporters in response to amino acid ingestion from baseline. The response before bed rest will be compared to after bed rest.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Reidy PT, Lindsay CC, McKenzie AI, Fry CS, Supiano MA, Marcus RL, LaStayo PC, Drummond MJ. Aging-related effects of bed rest followed by eccentric exercise rehabilitation on skeletal muscle macrophages and insulin sensitivity. Exp Gerontol. 2018 Jul 1;107:37-49. doi: 10.1016/j.exger.2017.07.001. Epub 2017 Jul 10. PMID 28705613
- [Derived] Carlin MB, Tanner RE, Agergaard J, Jalili T, McClain DA, Drummond MJ. Skeletal muscle Ras-related GTP binding B mRNA and protein expression is increased after essential amino acid ingestion in healthy humans. J Nutr. 2014 Sep;144(9):1409-14. doi: 10.3945/jn.114.196691. Epub 2014 Jul 23. PMID 25056691